CLINICAL TRIAL: NCT02450396
Title: Prospective Observational Study About Pregnancy and Medically Assisted Conception in Rare Diseases
Brief Title: Pregnancy and Medically Assisted Conception in Rare Diseases
Acronym: EGR2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: SNFMI (Unknown); SFR (Unknown); CRAT (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13.381bis
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Psoriatic Arthritis; Systemic Lupus Erythematosus; Antiphospholipid Syndrome; Sjogren Syndrome; Scleroderma; Myositis; Vasculitis; Mastocytosis; Various Autoimmune and/or Systemic and/or Rare Diseases
Keywords: Rare diseases; pregnancy; pregnancy,
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic; Lupus Erythematosus, Systemic; Antiphospholipid Syndrome; Sjogren's Syndrome; Scleroderma, Diffuse; Myositis; Vasculitis; Mastocytosis; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, cord blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Rare diseases frequently affect women of childbearing age. Pregnancy in these women has become less rare, but remains associated with high levels of complications. One obstacle to their optimal management during pregnancy is that there are no prospective studies of pregnancy during rare diseases and several connective tissue diseases. As a consequence, the management of these pregnancies is non-standardised in terms of treatment, monitoring (frequency of consultations, laboratory tests and ultrasound), and organisation of care.

Moreover, although these women (all diseases combined) are frequently exposed to medications potentially incompatible with pregnancy, little is known about the frequency of these exposures and especially their consequences to mother and child.

For these reasons, researchers and clinicians from different specialties created an interdisciplinary research group on pregnancy and rare diseases (GR2), intended to improve the management of these patients' pregnancies. Using a single computer server, the investigators plan to set up a large prospective study of pregnancies in patients with rare diseases: various forms of myositis, lupus, antiphospholipid syndrome, Sjogren syndrome, scleroderma, and inflammatory rheumatic diseases. The investigators objective is to analyse the complications of pregnancies in women with rare diseases and then to improve their management and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Woman with a rare and/or systemic disease
* Pregnancy confirmed by a positive beta-HCG assay or an obstetric ultrasound OR medically assisted conception procedure
* Patient agreed to participate

Exclusion Criteria:

* Adults under guardianship
* People hospitalised without their consent and not protected by the law
* Persons deprived of their liberty

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Woman with a rare and/or systemic disease Pregnancy confirmed by a positive beta-HCG assay or an obstetric ultrasound OR medically assisted conception procedure
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
"good" obstetric outcome | 35 week gestation until 1 year Post Partum
  It's a composite outcome . A pregnancy with no severe maternal complication (by the Epimoms* definition), live birth after 35 weeks' gestation, a birth weight >10th percentile of the general population and no infections (maternal and infant) during pregnancy and first year of follow up, respectively

SECONDARY OUTCOMES:
Define the best therapeutic management strategies | 2 years
  About the organisation of care (analysis of the effect on outcome of the number of ultrasound examinations and clinician visits, and the systematic planning of delivery)
Conduct pharmacoepidemiologic studies | 2 years
  Analyse the frequency of exposure to various medications (immunosuppressors, biological therapy, corticosteroids) and their maternal and fetal consequences (e.g., infectious complications).
Analyse the frequency of exposure to various medications (immunosuppressors, biological therapy, corticosteroids) and their maternal and fetal consequences (e.g., infectious complications). | 9 months
  Within an existing collection with (1) samples taken during the first trimester of pregnancy to analyse markers that might predict subsequent obstetric complications (cytokines, growth factors, enzymes) (2) with cord blood samples (which will, in particular, enable immunological and pharmacological analyses).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Costedoat-Chalumeau, PhD, Principal Investigator — Hôpital Cochin
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Derived] Dernoncourt A, Guettrot-Imbert G, Sentilhes L, Besse MC, Molto A, Queyrel-Moranne V, Besnerais ML, Lazaro E, Tieulie N, Richez C, Hachulla E, Sarrot-Reynauld F, Leroux G, Orquevaux P, London J, Sailler L, Souchaud-Debouverie O, Smets P, Godeau B, Pannier E, Murarasu A, Berezne A, Goulenok T, Morel N, Mouthon L, Duhaut P, Guern VL, Costedoat-Chalumeau N; Gr2 Study Group. Safety of Fertility Treatments in Women With Systemic Lupus Erythematosus: Data From a Prospective Population-Based Study. BJOG. 2025 Apr;132(5):614-624. doi: 10.1111/1471-0528.18050. Epub 2024 Dec 19. PMID 39702994
- [Derived] Alle G, Guettrot-Imbert G, Larosa M, Murarasu A, Lazaro E, Morel N, Orquevaux P, Sailler L, Queyrel V, Hachulla E, Sarrot Reynauld F, Perard L, Berezne A, Morati-Hafsaoui C, Chauvet E, Richez C, Goulenok T, London J, Molto A, Urbanski G, Le Besnerais M, Langlois V, Leroux G, Souchaud-Debouverie O, Roussin CL, Poindron V, Blanchet B, Pannier E, Sentilhes L, Mouthon L, Le Guern V, Costedoat-Chalumeau N; GR2 Study Group. Hydroxychloroquine levels in pregnancy and materno-fetal outcomes in systemic lupus erythematosus patients. Rheumatology (Oxford). 2025 Mar 1;64(3):1225-1233. doi: 10.1093/rheumatology/keae302. PMID 38837707
- [Derived] Murarasu A, Guettrot-Imbert G, Le Guern V, Yelnik C, Queyrel V, Schleinitz N, Ferreira-Maldent N, Diot E, Urbanski G, Pannier E, Lazaro E, Souchaud-Debouverie O, Orquevaux P, Belhomme N, Morel N, Chauvet E, Maurier F, Le Besnerais M, Abisror N, Goulenok T, Sarrot-Reynauld F, Deroux A, Pasquier E, de Moreuil C, Bezanahary H, Perard L, Limal N, Langlois V, Calas A, Godeau B, Lavigne C, Hachulla E, Cohen F, Benhamou Y, Raffray L, de Menthon M, Tieulie N, Poindron V, Mouthon L, Larosa M, Elefant E, Sentilhes L, Molto A, Deneux-Tharaux C, Costedoat-Chalumeau N; GR2 Study Group. Characterisation of a high-risk profile for maternal thrombotic and severe haemorrhagic complications in pregnant women with antiphospholipid syndrome in France (GR2): a multicentre, prospective, observational study. Lancet Rheumatol. 2022 Dec;4(12):e842-e852. doi: 10.1016/S2665-9913(22)00308-3. Epub 2022 Nov 24. PMID 38261392
- [Derived] Larosa M, Le Guern V, Guettrot-Imbert G, Morel N, Abisror N, Morati-Hafsaoui C, Orquevaux P, Diot E, Doria A, Sarrot-Reynauld F, Limal N, Queyrel V, Souchaud-Debouverie O, Sailler L, Le Besnerais M, Goulenok T, Molto A, Pannier-Metzger E, Sentilhes L, Mouthon L, Lazaro E, Costedoat-Chalumeau N; GR2 Group. Evaluation of lupus anticoagulant, damage, and remission as predictors of pregnancy complications in systemic lupus erythematosus: the French GR2 study. Rheumatology (Oxford). 2022 Aug 30;61(9):3657-3666. doi: 10.1093/rheumatology/keab943. PMID 35015828